CLINICAL TRIAL: NCT03811925
Title: Local and Systemic Vascular Function Following Drug Coated Balloon vs. Stenting in the Superficial Femoral Artery
Brief Title: SFA TReatment and vAscular Functions
Acronym: STRAtiFy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Fadi Al-Rashid, Principal Investigator, University Hospital, Essen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STRAtiFy_CR
Record Dates: First submitted 2019-01-16; First posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Peripheral Arterial Disease; Claudication, Intermittent
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB (Other)
  Interventions: Procedure: Angioplasty and drug coated balloon of the superficial femoral artery (SFA)
- Stenting (Other)
  Interventions: Procedure: Angioplasty and stenting of the superficial femoral artery (SFA)

INTERVENTIONS:
Procedure: Angioplasty and drug coated balloon of the superficial femoral artery (SFA) — In case of drug coated balloon (DCB) there should be always a predilation of the lesion with a predefined ballon (180 sec, Passeo-18). Thus, no direct DCB will be conducted. All DCB lengths (40mm to 200 mm) and Diameters (3mm to 7mm) are eligible for the Trial as long as used in the superficial femoral artery (SFA)
  Arms: DCB
Procedure: Angioplasty and stenting of the superficial femoral artery (SFA) — In case of stent application there should be always a predilation of the lesion with a predefined ballon (180 sec, Passeo-18). In case of stenting there should be a strong effect on vasomotion of the treated vessel area. All Stent lengths (40mm to 200 mm) and Diameters (5mm to 7mm) are eligible for the trial as long as used in the superficial femoral artery (SFA)
  Arms: Stenting

SUMMARY:
Endovascular treatment of the superficial femoral artery has a high initial success rate, but restenosis occurs in up to 60% of cases. While restoration of tissue perfusion is achieved, interventional strategies affect endothelial function. Endothelial dysfunction is the pathophysiologic principle involved in the initiation and progression of arteriosclerosis.

The aim of this study is to determine the impact of endovascular strategies in the superficial femoral artery on local and systemic endothelial and vascular function.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic, symptomatic lower limb ischemia as defined by Rutherford 2, 3, 4, or 5
* Planed peripheral intervention TASC A-C
* Subject must be between 40 and 85 years old
* Female of childbearing potential must have a negative pregnancy test within 10 days prior to index procedure and utilize reliable birth control until completion of the 12-month angiographic evaluation
* Guidewire must cross lesion(s) within the true lumen, without a relevant sub-intimal course
* Vessel diameter ≥3.0 mm and ≤6.0 mm
* Willing to comply with the specified follow-up evaluation
* Written informed consent prior to any study procedures

Exclusion Criteria:

* Lesions TASC D
* Angiographic evidence of thrombus within target vessel
* Thrombolysis within 72 hours prior to the index procedure
* Aneurysm in the femoral artery or popliteal artery
* Concomitant hepatic insufficiency, deep venous thrombus, coagulation disorder or receiving immunosuppressant therapy
* Unstable angina pectoris at the time of the enrollment
* Recent myocardial infarction or stroke < 30 days prior to the index procedure
* Life expectancy less than 12 months
* Septicemia at the time of enrollment
* Known or suspected active infection at the time of the index procedure, excluding an infection of a lower extremity wound of the target limb
* Known or suspected allergies or contraindications to aspirin, clopidogrel or heparin
* Presence of other hemodynamically significant outflow lesions in the target limb requiring a planned surgical intervention or endovascular procedure within 30 days after the index procedure

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
local endothelial function | 6 months Follow Up
  Change of endothelial function, assessed by the change in the vasodilatative reserve of the femoral artery (flow-mediated dilation = FMD)

SECONDARY OUTCOMES:
Systemic endothelial function | 6 months Follow Up
  1.Change of endothelial function, assessed by the change in the vasodilatative reserve of the brachial artery (flow-mediated dilation = FMD)
Vessel stiffness | 6 months Follow Up
  Vascular stiffness determined through pulse wave velocity (PWV)
Primary patency | 6 months Follow Up
  determined through doppler ultrasound
target lesion revascularization | 6 months Follow Up
  freedom from Target Lesion Revascularization (FTLR) is defined as the Need for percutaneous or interventional revascularization
ABI (Ankle Brachial Index) | 6 months Follow Up
  Ankle Brachial Index assessed by Doppler

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No